CLINICAL TRIAL: NCT02601664
Title: Randomized-controlled Trial of a Combined vs. Conventional Percutaneous Intervention for Near-Infrared Spectroscopy Defined High-Risk Native Coronary Artery Lesions
Acronym: CONCERTO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to lack of eligible patients.
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director of Cardiac Catheterization Laboratories, Professor of Medicine, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-083
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Arteriosclerosis; Near-infrared Spectroscopy; Peri-procedural Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Arteriosclerosis; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined Intervention (Active Comparator): Combined intervention: pre-PCI intracoronary vasodilator and glycoprotein IIb/IIIa inhibitor administration, use of an EPD if technically feasible, and complete coverage of the lipid core plaque, if technically feasible
  Interventions: Procedure: Combined Intervention
- Conventional PCI (Active Comparator): Conventional PCI
  Interventions: Procedure: Conventional PCI

INTERVENTIONS:
Procedure: Combined Intervention — pre-PCI intracoronary vasodilator administration and glycoprotein IIb/IIIa inhibitor administration, use of an embolization protection device if technically feasible, and complete coverage of the lipid core plaque, if technically feasible
  Arms: Combined Intervention
Procedure: Conventional PCI — Conventional PCI
  Arms: Conventional PCI

SUMMARY:
Design: Single center, single-blind randomized controlled trial of patients with high risk native coronary artery lesions (defined as ≥2 contiguous yellow blocks on the block chemogram) requiring clinically indicated percutaneous coronary intervention. Patients will be randomized to either a combined intervention or conventional PCI. Cardiac biomarker measurements will be performed before PCI and 18-24 hours later.

Treatment: Combined intervention consisting of pre-PCI intracoronary vasodilator and glycoprotein IIb/IIIa inhibitor administration, use of an EPD if technically feasible, and complete coverage of the lipid core plaque, if technically feasible.

Control: Conventional PCI. Duration: 30 days follow-up. The primary trial objective is to compare the incidence and size of periprocedural MI, as assessed by the peak post-PCI troponin distribution in the two study groups.

The secondary endpoints are: (1) Reduction in the incidence of >3x and >10x upper limit of normal increase in CK-MB. (2) Reduction in the incidence of slow flow/no-reflow post PCI. (3) Lower incidence of major adverse cardiac events, defined as the composite of death, acute coronary syndrome, or coronary revascularization) during 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Willing and able to provide informed consent and able to comply with study procedures and follow-up.
3. Undergoing a clinically indicated left heart coronary catheterization
4. Need PCI of a high-risk native coronary artery lesion. High-risk lesions will be defined as lesions with ≥2 contiguous yellow blocks on block chemogram.

Exclusion Criteria:

1. Coexisting conditions that limit life expectancy to less than 30-days or that could affect the patient's compliance with the protocol.
2. Positive pregnancy test or breast-feeding.
3. High risk for bleeding.
4. Subject is currently, or within the 30 preceding days, participating in a device or pharmaceutical treatment protocol.
5. Clinical presentation with ST-segment elevation MI.
6. Persistent (>10 minutes) hypotension (systolic blood pressure <90 mmHg)
7. Need for revascularization of multiple lesions during the index PCI.
8. Unprotected left main (>50%) or equivalent left main disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Reduction of the incidence and size of periprocedural MI, as assessed by the peak post-PCI troponin distribution | 18-24 hours post-procedure

SECONDARY OUTCOMES:
Reduction in the incidence of >3x and >10x upper limit of normal increase in CK-MB | 18-24 hours post-procedure
Reduction in the incidence of slow flow/no-reflow post PCI | 2-3 hours after
Lower incidence of major adverse cardiac events, defined as the composite of death, acute coronary syndrome, or coronary revascularization) during 30-day follow-up | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Study Chair — North Texas Veterans Healthcare System

REFERENCES:
- [Background] Brilakis ES, Abdel-Karim AR, Papayannis AC, Michael TT, Rangan BV, Johnson JL, Banerjee S. Embolic protection device utilization during stenting of native coronary artery lesions with large lipid core plaques as detected by near-infrared spectroscopy. Catheter Cardiovasc Interv. 2012 Dec 1;80(7):1157-62. doi: 10.1002/ccd.23507. Epub 2012 Apr 17. PMID 22511587
- [Background] Raghunathan D, Abdel-Karim AR, Papayannis AC, daSilva M, Jeroudi OM, Rangan BV, Banerjee S, Brilakis ES. Relation between the presence and extent of coronary lipid core plaques detected by near-infrared spectroscopy with postpercutaneous coronary intervention myocardial infarction. Am J Cardiol. 2011 Jun 1;107(11):1613-8. doi: 10.1016/j.amjcard.2011.01.044. PMID 21575750
- [Background] Patel VG, Brayton KM, Mintz GS, Maehara A, Banerjee S, Brilakis ES. Intracoronary and noninvasive imaging for prediction of distal embolization and periprocedural myocardial infarction during native coronary artery percutaneous intervention. Circ Cardiovasc Imaging. 2013 Nov;6(6):1102-14. doi: 10.1161/CIRCIMAGING.113.000448. No abstract available. PMID 24254480
- [Background] Stone GW, Maehara A, Muller JE, Rizik DG, Shunk KA, Ben-Yehuda O, Genereux P, Dressler O, Parvataneni R, Madden S, Shah P, Brilakis ES, Kini AS; CANARY Investigators. Plaque Characterization to Inform the Prediction and Prevention of Periprocedural Myocardial Infarction During Percutaneous Coronary Intervention: The CANARY Trial (Coronary Assessment by Near-infrared of Atherosclerotic Rupture-prone Yellow). JACC Cardiovasc Interv. 2015 Jun;8(7):927-36. doi: 10.1016/j.jcin.2015.01.032. Epub 2015 May 20. PMID 26003018
- [Background] Erlinge D, Harnek J, Goncalves I, Gotberg M, Muller JE, Madder RD. Coronary liposuction during percutaneous coronary intervention: evidence by near-infrared spectroscopy that aspiration reduces culprit lesion lipid content prior to stent placement. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):316-24. doi: 10.1093/ehjci/jeu180. Epub 2014 Sep 28. PMID 25266075